CLINICAL TRIAL: NCT07006948
Title: Multicenter Validation Study on the Effectiveness of a Machine-Assisted System for Early Screening of Autism
Brief Title: Multicenter Validation Study on Autism Screening Using a Machine-assisted System
Status: Not yet recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Harbin Institute of Technology, Shenzhen (Unknown); Kunshan City Maternal and Child Health (Other); Hefei First People's Hospital (Unknown); Ningbo Women & Children's Hospital (Other); Xiamen Children's Hospital (Other); Chengdu Women's and Children's Central Hospital (Other); Liuzhou Maternity and Child Healthcare Hospital (Other); Xian Children's Hospital (Other Government); Dehong People's Hospital (Unknown); The Sixth Affiliated Hospital of Harbin Medical University (Unknown)
Responsible Party: Sponsor
Other Study IDs: AI multicenter
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder; Early Developmental Impairment; Language Development Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Language Development Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ASD group: This group includes toddlers diagnosed with autism spectrum disorder aged between 1.5 to 2.5 years old.
  Interventions: Diagnostic Test: Autism Diagnostic Observation Schedule, the 2nd edition(ADOS-2); Diagnostic Test: Griffiths Developmental Scales, Chinese edition(GDS-C)
- GDD group: This group includes toddlers diagnosed with global development disorder aged between 1.5 to 2.5 years old.
  Interventions: Diagnostic Test: Griffiths Developmental Scales, Chinese edition(GDS-C)
- LD group: This group includes toddlers diagnosed with language disorder aged between 1.5 to 2.5 years old.
  Interventions: Diagnostic Test: Griffiths Developmental Scales, Chinese edition(GDS-C)
- TD group: This group includes typically developing toddlers aged between 1.5 to 2.5 years old.
  Interventions: Diagnostic Test: Griffiths Developmental Scales, Chinese edition(GDS-C)

INTERVENTIONS:
Diagnostic Test: Autism Diagnostic Observation Schedule, the 2nd edition(ADOS-2) — The toddlers diagnosed with ASD will receive the ADOS-2 evaluation to confirm the diagnosis.
  Groups: ASD group
Diagnostic Test: Griffiths Developmental Scales, Chinese edition(GDS-C) — The toddlers diagnosed with ASD, GDD, LD, and typically developing will receive the GDS-C evaluation to confirm the diagnosis.

SUMMARY:
The goal of this observational study is to assess the effectiveness of a machine-assisted system for early screening of autism. The main questions it aims to answer are:

* Does the machine-assisted system including 5 main behavioral paradigms identify toddlers with autism from those with other neurodevelopmental disorders and typical development?
* Are there any differences in the early symptoms of autism among toddlers over the whole mainland China? Participants will receive some developmental and social communicational evaluations for clinical diagnoses. They will also receive the behavior evaluations of the machine-assisted system. The above evaluations will be performed just once.

DETAILED DESCRIPTION:
The current study is a diagnostic accuracy study. In total, 1000 Toddlers with autism spectrum disorder, global developmental delay, language disorder, and typical development (n=250 for each group) will be recruited in this study. The gold standard of the diagnosis of autism spectrum disorder will be the clinical diagnosis from developmental and behavioral pediatricians, and the diagnoses will be confirmed by Autism Diagnostic Observation Schedule-2nd edition and Griffiths Development Scales-Chinese edition(GDS-C). The diagnostic accuracy of the machine-assisted system for early screening of autism will be evaluated.

ELIGIBILITY:
ASD group：

Inclusion Criteria:

1. Children diagnosed with ASD according to a clinical judgement based on the criteria of ASD in DSM-5 and further confirmed with ADOS-2;
2. Ages 1.5-2.5 years;
3. Parents/caregivers understand the content of the study and agree to participate in.

GDD group：

Inclusion Criteria:

1. Age 1.5-2.5 years, gestational age 37-42 weeks, birth weight 2500-4000g;
2. Clinically diagnosed with GDD (Global Developmental Delay) according to the DSM-V diagnostic criteria, with a Griffiths Development Scales-Chinese edition(GDS-C) assessment showing a Developmental Quotient (DQ) ≤75 in two or more domains;
3. Those who did not meet the initial screening positivity criteria for ASD (Autism Spectrum Disorder) using M-CHAT-R/F.

LD group：

Inclusion Criteria:

1. Age 1.5-2.5 years, gestational age 37-42 weeks, birth weight 2500-4000 g;
2. Clinically diagnosed with LD (Language Disorder) according to the DSM-V diagnostic criteria, with a Developmental Quotient (DQ) ≤75 in the language domain of the Griffiths Development Scales-Chinese edition(GDS-C) and DQ >75 in all other domains;
3. Those who did not meet the initial screening positivity criteria for ASD (Autism Spectrum Disorder) assessed by M-CHAT-R/F

Exclusion Criteria for ASD, GDD, and LD groups:

1. Rett Syndrome, Fragile X Syndrome, Angelman Syndrome, Prader-Willi Syndrome, tuberous sclerosis, and other syndromes caused by known genetic defects or inherited metabolic diseases;
2. Children with brain injuries, specific chronic or congenital diseases.
3. The gestational age is less than 37 weeks, or the birth weight is lower than 2500g.

TD group：

Inclusion Criteria:

1. Healthy, typically developing toddlers aged 1.5-2.5 years ;
2. gestational age of 37-42 weeks, birth weight of 2500-4000 g;
3. Developmental Quotients(DQs) are greater than 75 in all domains of theGriffiths Development Scales-Chinese edition(GDS-C);
4. Screened negative by M-CHAT-R/F screening for autism spectrum disorder (ASD).

Exclusion Criteria:

Children with neurodevelopmental disorders (e.g., developmental delay, language impairment), neurological conditions (e.g., epilepsy, tuberous sclerosis), or other severe chronic diseases were excluded.

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The diagnostic accuracy study will be performed in children with ASD, GDD, LD, and healthy, typically developing children aged between 1.5 to 2.5 years old.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
Total Score of 5 main social behaviors | The assessment will be performed during 1.5 to 2.5 years old.
  The 5 main social behaviors include Response to name, Response to instructions, Joint attention, request by pointing, and free play. Scores of the 5 scenes range from 0 to 4, and the total score ranges from 0 to 16. Higher score indicates better social skills. Subjects' behaviors will be scored both by investigators and the machine-assisted system.
Clinical diagnoses | The diagnoses will be made during 1.5 to 2.5 years old.
  The clinical diagnoses of autism spectrum disorder (ASD), global developmental delay (GDD), and language disorder (LD) will be made according to the standard of DSM-5. The diagnosis of ASD will be confirmed by The Modified Checklist for Autism in Toddlers, Revised with Follow-Up (M-CHAT-R/F) and Autism Diagnostic Observation Schedule, the 2nd edition (ADOS-2). The diagnoses of GDD and LD will be confirmed by Griffiths Development Scales-Chinese edition (GDS-C). Subjects in TD group will also receive assessments of M-CHAT-R/F, (negative) and GDS-C (DQs>75).
Scores of Autism Diagnostic Observation Schedule-2nd edition(ADOS-2) | The assessment will be performed during 1.5 to 2.5 years old.
  The scores of social affect and restricted repetitive behaviors and the comparison score of ADOS-2 will be used for confirming the clinical diagnosis of autism spectrum disorder(ASD). The minimum and maximum scores of ADOS-2 are 0 and 28, and the comparison score of ADOS-2 ranges from 1 to 10, in which higher scores mean a worse outcome.
development quotient development quotient Development quotients (DQs) of Griffiths Developmental Scales-Chinese edition(GDS-C) | The assessment will be performed during 1.5 to 2.5 years old.
  DQs of Griffiths Development Scales-Chinese edition(GDS-C) will be used for confirming the diagnoses of global developmental delay(GDD) and language disorder(LD), also be used to evaluate the development level of typically developing toddlers. The average scores of DQ in different domains are 100, and the standard deviations are 15. The DQ lower than 70(including 70) means lower than normal.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Xu, Principal Investigator — Children's Hospital of Fudan University
Locations (10):
- China (10):
  - Hefei First People's Hospital, Hefei, Anhui
  - Xiamen Children's Hospital, Xiamen, Fujian
  - Liuzhou Maternity and child Healthcare Hospital, Liuchow, Guangxi
  - The Sixth Affiliated Hospital of Harbin Medical University, Harbin, Helongjiang
  - Kunshan Maternal and Child Health Care Hospital, Kunshan, Jiangsu
  - Xi'an Children's Hospital, Xi'an, Shaanxi
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Dehong People's Hospital, Dehong, Yunnan
  - Ningbo Women and Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No